CLINICAL TRIAL: NCT01914536
Title: A Natural History Study of Adult Onset Pompe Disease Using Muscle MRI
Acronym: POMPE 2013
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: IIBSP-POM-2013-46
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Pompe Disease
Keywords: POMPE; Glycogenosis type II; Acid maltase deficiency
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood an urine samples will be obtained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pompe patients: Adult onset pompe patients being or not treated with enzyme therapy replacement

SUMMARY:
This project is an observational prospective study in which patients affected by an adult onset Pompe disease will be followed-up during three years using different clinical, analytical and radiological tests in order to know which is the natural history of the disease and which is the impact that treatment with recombinant enzyme has in the progression of the disease.

DETAILED DESCRIPTION:
Study aim:

The principal objective of the study is to find biomarkers that quantify the natural progression of the disease and to know if they are useful to determine the improvement or lack of impairment of the disease in response to Enzyme Replacement Therapy (ERT).

Study design:

A single center observational prospective study.

Patients:

Patients with adult onset POMPE disease (onset of symptoms after two years old) and molecular diagnosis confirming the disease are eligible

Methods:

Clinical information will be obtained according to a pre-defined protocol including six visits: screening visit, baseline, 6 month, 12 month, 24 month and 36 month.

In each visit we will perform the following tests: clinical assessment (including interview with patients, quality of live questionnaires, timed tests and assessment of muscle balance using a myometer), analytical tests (blood and urine tests), cardiac test (Electrocardiogram (ECG) and cardiac echography), respiratory assessment (using spirometer) and skeletal muscle imaging (Muscle MRI).

All data collect will be introduced in a database and afterwards statistically analyzed.

Expected results:

We expect to find a biomarker useful to follow-up the progression of Pompe disease. This biomarker has to be sensitive to the changes that muscle function may have after treatment with ERT.

Funding:

This project is funded by Genzyme, a Sanofi company

ELIGIBILITY:
Inclusion Criteria:

* Pompe disease confirmed using genetic study
* Onset of symptoms more than 2 years old
* To be able to come to the hospital and follow all the visits
* Patients with respiratory involvement are welcomed

Exclusion Criteria:

* Patients unable to perform a MRI (respiratory problems can be solved using mechanical ventilation)

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult onset Pompe Patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Changes in muscle atrophy using muscle MRI in patients with adult onset Pompe disease | baseline, 6 months, one year, two years and three years
  To know the natural progression of the disease regarding muscle atrophy measured using muscle MRI during a period of three years.

SECONDARY OUTCOMES:
Muscle strength | baseline, 6 months, one year, two years and three years
  To study progression of muscle weakness using manual and informatic devices as myometry. We will compare clinical progression with Muscle MRI results.
Micro RNA study | baseline, 6 months, one year, two years and three years
  We will obtain blood samples of all the patients to study the microRNA profile and different time points

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Díaz Manera, MD PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Isabel Illa, MD pHD, Study Director — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu iSant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Carrasco-Rozas A, Fernandez-Simon E, Lleixa MC, Belmonte I, Pedrosa-Hernandez I, Montiel-Morillo E, Nunez-Peralta C, Llauger Rossello J, Segovia S, De Luna N, Suarez-Calvet X, Illa I; Pompe Spanish Study group; Diaz-Manera J, Gallardo E. Identification of serum microRNAs as potential biomarkers in Pompe disease. Ann Clin Transl Neurol. 2019 Jul;6(7):1214-1224. doi: 10.1002/acn3.50800. Epub 2019 Jun 12. PMID 31353854